CLINICAL TRIAL: NCT07282769
Title: Once Weekly Semaglutide Treatment of Trichotillomania: An Open-Label Study
Brief Title: Semaglutide (Wegovy) Treatment for Trichotillomania
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-1571
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Trichotillomania (Hair-Pulling Disorder); Trichotillomania; Hair Pulling Disorder; Hair Pulling; Hair-Pulling Disorder
Keywords: trichotillomania; hair pulling
MeSH Terms: conditions — Trichotillomania | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Semaglutide (Wegovy) (Experimental): Participants will receive semaglutide (Wegovy) weekly for 8 weeks.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — All participants in the study will receive semaglutide (Wegovy).
  Other Names: Wegovy

SUMMARY:
This research study is testing the effectiveness and safety of semaglutide (Wegovy) in people with trichotillomania, also known as hair-pulling disorder.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy and safety of semaglutide in individuals with trichotillomania. The hypothesis to be tested is that semaglutide will reduce urges to pull hair and pulling behavior and will be well tolerated in participants with trichotillomania. The proposed study will provide needed pilot data on the treatment of a disabling disorder that currently lacks available options for pharmacological treatment.

The investigators will conduct an open-label pharmacotherapy trial in 10 individuals with trichotillomania. Participants with trichotillomania will be started and continued on medication during an 8-week treatment phase. The study will be the first to use a once weekly Glucagon-like peptide 1 (GLP-1) receptor agonist pharmacological intervention to target urges in trichotillomania and thereby has the potential to set a new standard of care for a range of compulsive behaviors.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-75;
2. Diagnosis of current trichotillomania based on DSM-5 criteria and confirmed using the clinician-administered MIDI (13);
3. Hair pulling daily with urges to pull as the trigger in >50% of the episodes of pulling;
4. Women of childbearing age are required to have a negative result on a beta-human chorionic gonadotropin pregnancy test;
5. Women of childbearing potential utilizing a medically accepted form of contraception defined as double barrier, oral contraceptive, injectable contraceptive, implantable contraceptive devices, and abstinence

Exclusion Criteria:

1. Infrequent pulling (i.e. less than daily) or automatic pulling (i.e. no urges to pull);
2. Unstable medical illness or clinically significant abnormalities on laboratory tests, EKG, or physical examination at screen as determined by the investigator;
3. History of seizures;
4. Myocardial infarction within 6 months;
5. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
6. A need for medication other than semaglutide with possible psychotropic effects or unfavorable interactions as determined by the investigator;
7. Clinically significant suicidality (defined by the Columbia Suicide-Severity Rating Scale);
8. Lifetime history of bipolar disorder type I or II, schizophrenia, or any psychotic disorder;
9. Current skin picking disorder;
10. Initiation of psychotherapy or behavior therapy within 3 months prior to study baseline;
11. Initiation of psychotropic medications within 3 months prior to study baseline (stable doses will be allowed);
12. Previous treatment with semaglutide;
13. Use of any weight loss medications;
14. Body mass index (BMI, calculated as weight in kilograms divided by height in meters squared) less than 23;
15. Past-year substance use disorder other than tobacco use disorder or mild cannabis use disorder;
16. Recent (30-day) use of illicit drugs except cannabis;
17. History of diabetes, and current medical or neurological illness precluding participation based on physician judgment;
18. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia 2A or 2B;
19. History of pancreatitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
NIMH Trichotillomania Severity Scale | From screening to 1 week after last dose of study drug
  Clinician-rated scale assessing trichotillomania symptom severity over the past week that will be administered at all visits. Total scores range from 0-20. Higher scores indicate greater severity.

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement and Severity Scales | From screening to 1 week after last dose of study drug
  Clinician-administered scale consisting of two reliable and valid 7-item Likert scales used to assess severity and change in clinical symptoms. The CGI-S will be used at screening and the CGI-I will be used at every visit after screening. the CGI-S ranges from 1 = "not ill at all" to 7 = "among the most extremely ill." The CGI-I scale ranges from 1 = "very much improved" to 7 = "very much worse."
Massachusetts General Hospital Hair Pulling Scale | From screening to 1 week after last dose of study drug
  A 7-item self-report measure assessing trichotillomania severity over the past week. Total scores range from 0-28. Greater scores indicate worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No